CLINICAL TRIAL: NCT00421330
Title: Endovascular Versus Transabdominal Treatment of the Abdominal Aortic Aneurysm: the Dutch Randomised Endovascular Aneurysm Management (DREAM-) Trial
Brief Title: Dutch Randomised Endovascular Aneurysm Management (DREAM-) Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00/144
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal aortic aneurysm; AAA; randomised controlled trial; Endovascular repair; conventional open repair
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OR (Active Comparator): Open Aneurysm Repair
  Interventions: Procedure: Open Aneurysm Repair
- EVAR (Experimental): Endovascular Aneurysm Repair
  Interventions: Procedure: Endovascular Aneurysm Repair

INTERVENTIONS:
Procedure: Open Aneurysm Repair
  Arms: OR
Procedure: Endovascular Aneurysm Repair
  Other Names: Excluder, Talent, Zenith, AneuRx
  Arms: EVAR

SUMMARY:
The purpose of this trial is to assess whether the new endovascular repair technique of the abdominal aortic aneurysm (AAA) is an adequate substitute of the conventional AAA repair.

DETAILED DESCRIPTION:
After the introduction of endovascular repair of abdominal aortic aneurysms (AAA), both benefits and drawbacks of this new technique have been reported. To assess whether the new technique is an adequate substitute of conventional AAA repair, a randomised study is required. The DREAM trial is a randomised multicenter trial enrolling patients eligible for elective treatment of infrarenal AAAs. The primary endpoint is combined operative mortality and morbidity. Secondary endpoints and additional assessments include event-free survival, quality of life,and costs.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic, infrarenal AAA that requires surgery
* Adequate infrarenal neck
* Other aortic-iliac anatomical configuration suitable for EVAR according to the criteria of the device to be used
* Patient having a life expectation of at least 2 years and cleared for transabdominal intervention
* Signed informed consent

Exclusion Criteria:

* ruptured AAA or symptomatic AAA, which requires emergency surgery
* maximum aneurysm diameter< 5.0 cm
* suprarenal AAA
* Inflammatory AAA (more than minimal wall thickening)
* infrarenal neck unsuitable for endovascular fixation or aortic-iliac anatomic configuration otherwise unsuitable for EVAR according to criteria of the device to be used
* bilateral retroperitoneal incision required for EVAR
* sacrifice of both hypogastric arteries required
* anatomical variations, i.e. horseshoe-kidney, arteries requiring reimplantation
* patient unsuitable for laparotomy
* administration of contrast agent not possible: proved, severe systemic reaction to contrast agent
* active infection present
* transplantation-patients
* limited life expectation due to other illness (< 2 year)
* non-iatrogenic bleeding diathesis
* connective tissue disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2000-11; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
combined operative mortality and morbidity | 5-8 years

SECONDARY OUTCOMES:
event free survival | 5-8 years
quality of life | 5-8 years
cost-effectiveness | 5-8 years

CONTACTS AND LOCATIONS:
Overall Officials: J D Blankensteijn, MD, PhD, Principal Investigator — Radboud University Nijmegen Mecial Center, The Netherlands

REFERENCES:
- [Result] Prinssen M, Buskens E, Blankensteijn JD. The Dutch Randomised Endovascular Aneurysm Management (DREAM) trial. Background, design and methods. J Cardiovasc Surg (Torino). 2002 Jun;43(3):379-84. PMID 12055570
- [Result] Prinssen M, Verhoeven EL, Buth J, Cuypers PW, van Sambeek MR, Balm R, Buskens E, Grobbee DE, Blankensteijn JD; Dutch Randomized Endovascular Aneurysm Management (DREAM)Trial Group. A randomized trial comparing conventional and endovascular repair of abdominal aortic aneurysms. N Engl J Med. 2004 Oct 14;351(16):1607-18. doi: 10.1056/NEJMoa042002. PMID 15483279
- [Result] Prinssen M, Buskens E, Blankensteijn JD; DREAM trial participants. Quality of life endovascular and open AAA repair. Results of a randomised trial. Eur J Vasc Endovasc Surg. 2004 Feb;27(2):121-7. doi: 10.1016/j.ejvs.2003.11.006. PMID 14718892
- [Result] Prinssen M, Buskens E, Nolthenius RP, van Sterkenburg SM, Teijink JA, Blankensteijn JD. Sexual dysfunction after conventional and endovascular AAA repair: results of the DREAM trial. J Endovasc Ther. 2004 Dec;11(6):613-20. doi: 10.1583/04-1280R.1. PMID 15615551
- [Result] Blankensteijn JD, de Jong SE, Prinssen M, van der Ham AC, Buth J, van Sterkenburg SM, Verhagen HJ, Buskens E, Grobbee DE; Dutch Randomized Endovascular Aneurysm Management (DREAM) Trial Group. Two-year outcomes after conventional or endovascular repair of abdominal aortic aneurysms. N Engl J Med. 2005 Jun 9;352(23):2398-405. doi: 10.1056/NEJMoa051255. PMID 15944424
- [Derived] van Schaik TG, Yeung KK, Verhagen HJ, de Bruin JL, van Sambeek MRHM, Balm R, Zeebregts CJ, van Herwaarden JA, Blankensteijn JD; DREAM trial participants. Long-term survival and secondary procedures after open or endovascular repair of abdominal aortic aneurysms. J Vasc Surg. 2017 Nov;66(5):1379-1389. doi: 10.1016/j.jvs.2017.05.122. PMID 29061270
- [Derived] de Bruin JL, Baas AF, Heymans MW, Buimer MG, Prinssen M, Grobbee DE, Blankensteijn JD; DREAM Study Group. Statin therapy is associated with improved survival after endovascular and open aneurysm repair. J Vasc Surg. 2014 Jan;59(1):39-44.e1. doi: 10.1016/j.jvs.2013.07.026. Epub 2013 Oct 18. PMID 24144736
- [Derived] de Bruin JL, Vervloet MG, Buimer MG, Baas AF, Prinssen M, Blankensteijn JD; DREAM Study Group. Renal function 5 years after open and endovascular aortic aneurysm repair from a randomized trial. Br J Surg. 2013 Oct;100(11):1465-70. doi: 10.1002/bjs.9280. PMID 24037566
- [Derived] De Bruin JL, Baas AF, Buth J, Prinssen M, Verhoeven EL, Cuypers PW, van Sambeek MR, Balm R, Grobbee DE, Blankensteijn JD; DREAM Study Group. Long-term outcome of open or endovascular repair of abdominal aortic aneurysm. N Engl J Med. 2010 May 20;362(20):1881-9. doi: 10.1056/NEJMoa0909499. PMID 20484396